CLINICAL TRIAL: NCT00257413
Title: Safety and Efficacy Study of Transplantation of EPCs to Treat Idiopathic Pulmonary Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-007
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2005-11-22 (Estimated); Status verified 2003-12

CONDITIONS: Idiopathic Pulmonary Arterial Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension

INTERVENTIONS:
Procedure: Transplantation of autologous endothelial progenitor cells

SUMMARY:
Experimental data suggest that transplantation of endothelial progenitor cells (EPCs) attenuates monocrotaline-induced pulmonary hypertension in rats and dogs. In addition, clinical studies suggest that autogolous progenitor cells transplantation is feasible and safe in patients with ischemic disease. This study will investigate the feasibility, safety, and initial clinical outcome of intravenous infusion of autologous EPCs in patients with idiopathic pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic pulmonary arterial hypertension
* in New York Heart Association (NYHA) functional class II to III
* a mean pulmonary artery pressure more than 30 mmHg on right heart catheterization
* the ability to walk ≥50 m during a standardized 6-minute walk test.

Exclusion Criteria:

* Pulmonary hypertension as a result of heart disease, pulmonary disease, sleep-associated disorders, chronic thromboembolic disease, autoimmune or collagen vascular disease, HIV infection, liver disease, NYHA functional class IV, major bleeding requiring blood transfusion, diabetes, renal dysfunction, and evidence for malignant diseases were excluded

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: junzhu chen, MD, Study Chair — First Affiliated Hospital of Zhejiang University
Locations (1):
- Department of Cardiology, the First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Takahashi M, Nakamura T, Toba T, Kajiwara N, Kato H, Shimizu Y. Transplantation of endothelial progenitor cells into the lung to alleviate pulmonary hypertension in dogs. Tissue Eng. 2004 May-Jun;10(5-6):771-9. doi: 10.1089/1076327041348563. PMID 15265294
- [Derived] Wang XX, Zhang FR, Shang YP, Zhu JH, Xie XD, Tao QM, Zhu JH, Chen JZ. Transplantation of autologous endothelial progenitor cells may be beneficial in patients with idiopathic pulmonary arterial hypertension: a pilot randomized controlled trial. J Am Coll Cardiol. 2007 Apr 10;49(14):1566-71. doi: 10.1016/j.jacc.2006.12.037. Epub 2007 Mar 27. PMID 17418297